CLINICAL TRIAL: NCT00003541
Title: High Dose Combined Modality Therapy With Peripheral Blood Progenitor Cell Transplantation as Primary Treatment for Patients With Mantle Cell Lymphoma
Brief Title: Combination Chemotherapy, Radiation Therapy, and Peripheral Stem Cell Transplantation in Treating Patients With Stage III or Stage IV Mantle Cell Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 98-045; CDR0000066595 (Registry Identifier: PDQ (Physician Data Query)); NCI-H98-0021
Record Dates: First submitted 1999-11-01; First posted 2004-01-23 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2013-06

CONDITIONS: Lymphoma
Keywords: stage III mantle cell lymphoma; stage IV mantle cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Mantle-Cell | interventions — Filgrastim; VAP-cyclo protocol; Carboplatin; Cyclophosphamide; Doxorubicin; Etoposide; Ifosfamide; Prednisone; Vincristine; Peripheral Blood Stem Cell Transplantation; Radiotherapy

INTERVENTIONS:
Biological: filgrastim
Drug: CHOP regimen
Drug: carboplatin
Drug: cyclophosphamide
Drug: doxorubicin hydrochloride
Drug: etoposide
Drug: ifosfamide
Drug: prednisone
Drug: vincristine sulfate
Procedure: peripheral blood stem cell transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage cancer cells. Combining chemotherapy, radiation therapy, and peripheral stem cell transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more cancer cells.

PURPOSE: Phase I/II trial to study the effectiveness of combination chemotherapy, radiation therapy, and peripheral stem cell transplantation in treating patients who have stage III or stage IV mantle cell lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the response to a 8 week induction chemotherapy program consisting of cyclophosphamide, doxorubicin, vincristine, and prednisone (CHOP) in patients with mantle cell lymphoma. II. Evaluate the efficacy of ifosfamide, carboplatin, and etoposide (ICE) chemotherapy and filgrastim (G-CSF) for peripheral blood stem cell (PBSC) mobilization in this patient population. III. Evaluate the safety and efficacy of ICE followed by total body irradiation and high dose cyclophosphamide and etoposide in this patient population. IV. Assess the contamination of PBSCs by lymphoma cells following mobilization by chemotherapy and G-CSF in this patient population.

OUTLINE: Patients receive induction chemotherapy with cyclophosphamide IV, doxorubicin IV, and vincristine IV on day 1, oral prednisone daily on days 2-6, and filgrastim (G-CSF) subcutaneously daily on days 6-10. Treatment is repeated every 14 days for up to 4 courses. Patients receive consolidation chemotherapy with ifosfamide IV over 24 hours and carboplatin IV on day 2, etoposide IV daily on days 1-3, and G-CSF subcutaneously on days 5-12 for course 1, and on day 5 for course 2 and continuing through peripheral blood stem cell (PBSC) collection. Treatment is repeated every 14 days for 2 courses. Following PBSC collection, patients receive total body irradiation twice a day for 4 days plus etoposide IV over 72 hours on days -6, -5, and -4 and cyclophosphamide IV daily on days -3 and -2. PBSCs are infused on day 0. Patients receive G-CSF IV or subcutaneously twice a day beginning on day 1. Patients are followed every 3 months for 2 years, every 6 months for 3 years, and annually thereafter.

PROJECTED ACCRUAL: Approximately 14-24 patients will be accrued for this study within two years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed stage III or IV mantle cell lymphoma (diffuse, nodular, mantle zone, or blastic variants)

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Not specified Life expectancy: Not specified Hematopoietic: Not specified Hepatic: No chronic active or persistent hepatitis Bilirubin less than 2 mg/dL (unless history of Gilbert's disease) Renal: No history of chronic renal insufficiency Creatinine less than 1.5 mg/dL OR Creatinine clearance greater than 60 mL/min Cardiovascular: At least 6 months since myocardial infarction No unstable angina No cardiac arrhythmias other than chronic atrial fibrillation LVEF at least 50% Pulmonary: DLCO at least 50% Other: No medical illness that would preclude study treatment No uncontrolled infection No history of malignancy, other than curatively treated basal cell skin cancer or carcinoma in situ of the cervix Not pregnant or nursing Fertile patients must use effective contraception Not HIV positive

PRIOR CONCURRENT THERAPY: No prior therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 1998-06; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carol S. Portlock, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States